CLINICAL TRIAL: NCT04885140
Title: Effect of Feedback Health Education on Postoperative Rehabilitation of Patients With Lumbar Disc Herniation: a Cluster Randomized Trials
Brief Title: Effect of Feedback Health Education on Postoperative Rehabilitation of Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Hospital (Other)
Responsible Party: Principal Investigator, Fan Rong, Clinical Professor, Tianjin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Jiangsu College of Nursing
Record Dates: First submitted 2021-04-15; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Disc Herniation
Keywords: Feedback method; Health education; Functional exercise
MeSH Terms: conditions — Intervertebral Disc Displacement; Health Education

STUDY DESIGN:
Intervention Model Description: The methods were based on previous research on the feedback method of health education. A cluster randomized controlled trial design was used. From March 2019 to January 2020, patients who underwent spinal surgery at Tianjin Hospital were enrolled, and 76 met the inclusion criteria for lumbar disc disease (lumbar disc herniation, LDH). Patients were divided into an experimental group and a control group, with 38 patients in each group. Feedback-based health education was conducted for the experimental group, and routine health education was provided for the control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback-based health education health education and Routine health education (Experimental): Feedback-based health education:(1) Implementation of the feedback method includes information transmission, patient feedback, clarification and correction, and confirmation of understanding.① One day before surgery: Health education team members provided bedside one-on-one education for patients, 15-20 min per session, twice a day.
  ② One week after surgery: One-on-one education on rehabilitation exercise was conducted for the patients by the health education team members, 15-20 min per session, twice a day.
  ③ Two to four weeks after surgery: The health education group members guided the patients through functional rehabilitation exercises via WeChat. Each intervention lasted 20-30 min. The patients interacted once through WeChatB1, and their questions were answered at any time.
  ④ Five to 12 weeks after surgery: The health education group members guided patients through the functional rehabilitation exercises via WeChat.
  Interventions: Behavioral: Feedback-based health education
- Routine health education (Experimental): Routine health education:
  Routine health education was given to the patients, and the content of health education was the same as that of the experimental group, including the introduction of the disease, clinical manifestations, significance of examination, therapeutic principles of operative methods, psychological nursing, and postoperative rehabilitation exercise, etc. To verify the effect of health education by feedback method.
  Interventions: Behavioral: Routine health education

INTERVENTIONS:
Behavioral: Feedback-based health education — This study was approved by the Tianjin Hospital Ethics Committee, (2019082).The CONSORT 2010 statement: extension to cluster-randomised trials checklist.(Campbell et al., 2012) was used to guide reporting outcomes (File S1).Specific measures have been listed above.
  Arms: Feedback-based health education health education and Routine health education
Behavioral: Routine health education — Routine health education was given to the patients, and the content of health education was the same as that of the experimental group, including the introduction of the disease, clinical manifestations, significance of examination, therapeutic principles of operative methods, psychological nursing, and postoperative rehabilitation exercise, etc. To verify the effect of health education by feedback method.
  Arms: Routine health education

SUMMARY:
Aims and Objective: A theoretical model based on guided postoperative rehabilitation with feedback was developed for patients with lumbar intervertebral disc protrusion to explore the effects of feedback-based health education. Patients were assessed in terms of disease knowledge, general self-efficacy, medical behaviour, and the Oswestry disability index (ODI). During postoperative rehabilitation, nursing staff provided health education regarding lumbar intervertebral disc protrusion.

DETAILED DESCRIPTION:
Grouping method For the surgical treatment of lumbar intervertebral disc protrusion. The age of the included patients was greater than or equal to 18 years. Patients were cluster randomized by a coin toss into an experimental group that underwent spine surgery and a control group; 38 cases were included in each group for a total of 76 cases, and patients were assigned to the experimental and control groups in a 1:1 ratio, ensuring balance between groups. During implementation of the intervention, 1 patient in the control group voluntarily requested to withdraw from the study midway through the study, and the loss to follow-up rate was 2.6%. Finally, a total of 75 patients were included in this study, including 38 in the experimental group and 37 in the control group.

3 Test group

(1) Implementation of the feedback method includes information transmission, patient feedback, clarification and correction, and confirmation of understanding

① Conveying health information Medical terms were transformed into plain language so that patients could easily understand the health education content. The feedback method was used to explain the pathogenesis of LDH as protrusion or degeneration of the collodium supporting the lumbar spine and rupture of the cartilage protecting the lumbar spine. The protruding collodium compresses the nerve root, leading to pain in the back and leg.

* Patient feedback After a health message was delivered, the patient was asked to repeat the information back in his own words with the following question: To make sure I'm clear, could you repeat the pathogenesis for me?

  ③ Educator clarification and correction If the patient had mastered the relevant information, the health education session was ended. If the patient understood some or no information, the steps were repeated, and the educator continued to explain the concept to the patient but changed the way he or she expressed it.

  ④ Checking understanding Finally, open questions such as the following were used to confirm the patient's understanding: Do you have any other questions? The patients were then given a chance to sort out the health information.

  (2) Patients in the test group received health education according to the feedback method, and the intervention contents and time were as follows:

  ① One day before surgery: Health education team members provided bedside one-on-one education for patients, 15-20 min per session, twice a day. Health education manuals and other tools were used to explain information related to lumbar intervertebral disc herniation, including the pathogenesis of LDH, clinical manifestations, the significance of relevant examinations, the principle of surgical treatment, and the importance of exercising according to the guidance of doctors, to the patient. The main problem before LDH was pain in the waist and legs, so the patients were advised to take medication and taught how to take neurotropin, mecobalamine, Celebrex and other drugs.
* One week after surgery: One-on-one education on rehabilitation exercise was conducted for the patients by the health education team members, 15-20 min per session, twice a day.

Day of surgery: The main concerns of the patients were wound pain and axial rolling. After returning to the ward, the patients were taught about pain and the correct use of the analgesic pump.

One week after surgery: The main concerns of the patients were waist circumference and methods of rehabilitation exercise. Patients were instructed to perform straight leg raising exercises, ankle pump exercises and quad contraction exercises, 10~20 times/session, 3 sessions/day. If the patient understood the relevant knowledge and completed the rehabilitation exercise, the patient was affirmed and encouraged in the form of award certificates, and the "Best Cooperation Award", "Best Progress Award", "Most Confidence Award", "Three Good Fellow Award", etc., were used to enhance the patient's self-confidence, sense of honour and sense of achievement in rehabilitation exercise. In terms of discharge guidance, patients were told to go home and continue to perform functional exercise.

③ Two to four weeks after surgery: The main concerns of patients were functional exercise and daily life activities. The health education group members guided the patients through functional rehabilitation exercises via WeChat. Each intervention lasted 20-30 min. The patients interacted once through WeChatB1, and their questions were answered at any time. Patients were instructed to perform head lifting training in the prone position, a wood rolling exercise, walking training (waist-assisted) and supine hip flexion and knee flexion exercises, 5-10 min/session, 3 sessions/day. Patients were required to sign in after receiving new exercises and give feedback. Patients were required to "send a video of themselves performing functional exercise to the group", and the health education team members corrected any incorrect movement or frequency, answered their questions, and confirmed whether they understood until they had fully mastered the correct methods for the functional exercise. WeChat pushed small pieces of information twice via a link.

④ Five to 12 weeks after surgery: the main concerns of patients were functional exercise methods, such as five-point support, and other matters needing attention. The health education group members guided patients through the functional rehabilitation exercises via WeChat. Each intervention lasted 20~30 min, and WeChat was used for both sessions.

4 Control group: The patients underwent routine health education.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lumbar disc herniation Disease
* Must be able to Cooperate with research

Exclusion Criteria:

* Lumbar malignant tumors, lumbar tuberculosis and osteoporosis
* People with mental system diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
General data | Day 1
  The content includes general demographic and sociological data such as gender, age and education level, as well as basic information of diseases.
LDH knowledge questionnaire | Day 1 to week 12
  LDH knowledge questionnaire was prepared by Shi Yixin, with a total of 12 items. The questionnaire was scored by Likert 5, The minimum value is 1 point and the full score being 60 points. The higher the score, the better the patient's knowledge mastery. The content validity of knowledge questionnaire was 0.96 and Cronbach's α coefficient was 0.80.
General Self-Efficacy Scale | Day 1 to week 12
  In this study, Wang Caikang translated Chinese version of scale general self-efficacy scale consists of 10 entries, beliefs about individual when facing difficulties or problems, adopt Likert level 4 score, each item from "completely incorrect" to "completely correct" respectively in 1 ~ 4 points, The minimum value is 1 point and the maximum value is 40 points, the higher the score shows that the higher the self-efficacy of the patients. The content validity of the scale was 0.87 and Cronbach's α coefficient was 0.83.
Questionnaire on the compliance behaviour of LDH patients | Day 1 to week 12
  The questionnaire on compliance behavior of LDH patients was prepared by Shi Yixin, a researcher. The contents of the questionnaire included functional exercise, activities, diet, daily living, review, etc.The questionnaire adopts Likert 5 score, The minimum value is 1 point and the maximum value is 90 points. The higher the score, the better the compliance behavior of patients. The content validity of the questionnaire is 0.98, and Cronbach's α coefficient is 0.84.
Oswestry disability index (ODI) scale | Day 1 to week 12
  This scale is widely used in China and internationally, and in the field of spinal medicine, it is recognized as the gold standard for evaluating curative effects and function . The scale was compiled in 1980 by Fairbank and colleagues and has been revised since ; it was first used in China after it was adapted by Zheng Guangxin . The scale is used to evaluate the efficacy of surgical treatment and is an important reference index in patients with lumbar disease.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Rong Fan Rong, master, Principal Investigator — Tianjin Hospital
Locations (1):
- Jiangsu College of Nursing, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baretich M. National Quality Forum releases recommendations for safe practices. Biomed Instrum Technol. 2010 Jul-Aug;44(4):334-5. doi: 10.2345/0899-8205-44.4.334. No abstract available. PMID 20715962

DOCUMENTS (1):
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04885140/ICF_000.pdf